CLINICAL TRIAL: NCT05045248
Title: Efficacy of Apraclonidine Eye Drops in the Treatment of Ptosis Secondary to Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Johnny Salameh, Associate Professor, Department of Neurology, American University of Beirut Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2019-0027
Record Dates: First submitted 2021-08-29; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Myasthenia Gravis; Ocular Myasthenia Gravis
Keywords: myasthenia gravis; ocular myasthenia; apraclonidine
MeSH Terms: conditions — Myasthenia Gravis | interventions — apraclonidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients (Experimental): Each patient is administered 2 drops of Apraclonidine 0.5% solution to the most affected eye. Objective measurements of ptosis will be taken before drug administration and at 1, 5, 30, 60 minutes after drug administration in order to analyze any change in ptosis.
  Interventions: Drug: Apraclonidine Hcl 0.5% Oph Soln

INTERVENTIONS:
Drug: Apraclonidine Hcl 0.5% Oph Soln — Each patient is administered 2 drops of Apraclonidine 0.5% solution to the most affected eye
  Other Names: Iopidine 0.5%

SUMMARY:
This study is aimed at assessing the efficacy of Apraclonidine eye drops in the treatment of ptosis secondary to myasthenia gravis.

DETAILED DESCRIPTION:
The rationale behind using Apraclonidine is that it acts on Muller's muscle which is a sympathetic-innervated muscle. As such, this muscle is expected to be spared from the effects of the autoantibodies that attack the postsynaptic portion of the neuromuscular junction in myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older with a diagnosis of ocular or generalized myasthenia gravis with ocular involvement.

Exclusion Criteria:

* Patients receiving mono-amino-oxidase inhibitors.
* Patients with history of hypertension, cardiac, or cerebrovascular disease.
* Women with confirmed pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Change in palpebral fissure height (PF) | Before administration, at 1, 5, 30, and 60 minutes after administration
  Change in PF measurements
Change in marginal reflex distance-1 (MRD1) | Before administration, at 1, 5, 30, and 60 minutes after administration
  Change in MRD1 measurements
Change in marginal reflex distance-2 (MRD2) | Before administration, at 1, 5, 30, and 60 minutes after administration
  Change in MRD2 measurements
Change in levator function (LF) | Before administration, at 1, 5, 30, and 60 minutes after administration
  Change in LF measurements

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Salameh, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agha M, Ismail H, Sawaya R, Salameh J. Efficacy of apraclonidine eye drops in treating ptosis secondary to myasthenia gravis: A pilot clinical trial. Muscle Nerve. 2023 Aug;68(2):206-210. doi: 10.1002/mus.27851. Epub 2023 May 31. PMID 37259693